CLINICAL TRIAL: NCT05797922
Title: A Phase 1 Clinical Trial to Evaluate the Effect of Food on the Pharmacokinetics and Safety of DWP16001 After Administration in Healthy Adult Volunteers
Brief Title: To Evaluate the Effect of Food on the Safety and PK Characteristics of DWP16001 in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWP16001109
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP16001 to Group A (Experimental): Group A: Fasting in Period 1 / Fed in Period 2
  Interventions: Drug: DWP16001
- DWP16001 to Group B (Experimental): Group B: Fed in Period 1 / Fasting in Period 2
  Interventions: Drug: DWP16001

INTERVENTIONS:
Drug: DWP16001 — DWP16001 0.3mg
  Other Names: DWP16001 0.3mg

SUMMARY:
This study aims to evaluate the effect of food on the pharmacokinetics and safety of DWP16001 after oral administration.

DETAILED DESCRIPTION:
The study design is A randomized, Open-label, Oral, Single-dose, Two-way crossover study.

ELIGIBILITY:
Inclusion Criteria:

1. A person who has decided to participate voluntarily and agreed in writing prior to the screening procedure after understanding the detailed explanation of this clinical trial.
2. A person who is 19 years of age or more at the time of screening.
3. Those with a weight of 50.0 kg or more and a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less.

Exclusion Criteria:

1. A person who has a genetic problem such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
2. A person who has a history of gastrointestinal surgery/disease, such as Crohn's disease, ulcer, acute or chronic pancreatitis, which may affect the absorption of drug for clinical trials. (Except for simple appendectomy or hernia surgery)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-t of DWP16001 | 0 to 72 hours
  AUC0-t of DWP16001
Cmax of DWP16001 | 0 to 72 hours
  Cmax of DWP16001

CONTACTS AND LOCATIONS:
Overall Officials: Chungbuk National University Hospital, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Jungbuk, South Korea